CLINICAL TRIAL: NCT05322746
Title: Effects of Focal Vibrations on Neuropathic Pain in Diabetic Peripheral Neuropathy
Brief Title: Focal Vibrations and Neuropathic Pain in Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01225 Sameen Tahir
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Neuropathy; Diabetic Neuropathies
Keywords: Pain; Neuropathy; Diabetes
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetic Neuropathies; Pain; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Focal Muscle vibration will be apply to:
  1. Tibialis anterior
  2. The distal quadriceps
  3. Belly of the gastrocnemius/soleus muscles.
  4. Sinusoidal vibration intensity range 120 Hz.
  5. Each muscle will vibration for 10 minutes
  6. 10 minutes per muscle duration; total 30 minutes
  Interventions: Device: Focal muscle vibration
- Group B (Active Comparator): Focal Muscle vibration similar to Group A with following:
  Conventional Therapy TENS with pulse width 250ms, intensity 14Hz for 30 minutes
  Exercise therapy:
  Stretching Exercise to:
  1. Calf
  2. Hamstring
  3. Quadriceps
  Interventions: Device: Focal muscle vibration
- Group C (Active Comparator): TENS with pulse width 250ms, intensity 14Hz for 30 minutes
  Exercise therapy:
  Stretching Exercise to:
  1. Calf
  2. Hamstring
  3. Quadriceps
  Interventions: Device: Focal muscle vibration

INTERVENTIONS:
Device: Focal muscle vibration — Focal muscle vibration (FMV) defined as a technique that applies a vibratory stimulus to a specific muscle or its tendon using a mechanical device. FMV generates the Ia inputs as a consequence of the activation primary ending of the muscle spindle leading to alteration of corticospinal pathways results in activation of Ia inputs by FMV. The vibration of a specific muscle can increase the motor evoked potential, enhance the changes in corticospinal excitability and produces involuntary contraction in the vibrated muscle

SUMMARY:
Most of the literature found on whole body vibrations(WBV) instead of focal muscle vibrations (FMV) in diabetic peripheral neuropathy patients. The studies found on the effects of focal vibrations could not be generalised on the huge population of diabetes mellitus (DM) induced neuropathic pain because of small sample size and due to subordinate studies i.e, pilot studies done on the focal vibrations in which 3 different modes of vibrations is used without comparing with the control group. These studies are not much valuable in literature as well as for clinical purposes due to lack of control group. As mentioned in previous studies that better results achieved with the WBV on pain in diabetic peripheral neuropathyso that the hypothesis can be made that when FMV directly applies on the focal region that may influence the pain and/or peripheral neuropathy status.

DETAILED DESCRIPTION:
Diabetic neuropathy is the most common complication associated with diabetes mellitus, affecting approximately 50-70% of patients with diabetes. The prevalence of pain and of paraesthesia were 20% and 33% 10 years after diagnosis of diabetes mellitus (DM). DPN is the leading cause for disability due to foot ulceration and amputation and significantly lowers quality of life (QoL). Neuropathic pain is caused by a lesion or disease of the somatosensory system, including peripheral fibres (Aβ, Aδ and C fibres) and central neurons. Thus the prevalence of DPN and limitations of current studies make evident the need for future research.The study going to be taken with a large sample size, further testing the efficacy of FMV as a treatment for DPN and also check the detraining effects after discontinuation of therapy for 1 month so that the gaps in the literature can be full filled

ELIGIBILITY:
Inclusion Criteria:

* Diabetic type II patients.
* Score >12 at Leeds Assessment of Neuropathic Symptoms & Signs (LANSS)
* Diagnosis of diabetic peripheral neuropathy, using previous history, physical examination and vibration perception test of the patients
* Post diabetic duration of 10 years
* Patient with lower limb pain ranges from 3 to 5 on short form McGill pain

Exclusion Criteria:

* Lower extremity amputation
* Neuropathy other than diabetes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Short Form McGill Pain Questionnaire | 0 week
  Short Form McGill Pain Questionnaire is used to assess the non-neuropathic or neuropathic pain and describe the different qualities of pain and related symptoms. It has 0 to 10 scale, with 0 begin no pain and 10 begin worst pain.
Short Form McGill Pain Questionnaire | 4 weeks
  Short Form McGill Pain Questionnaire is used to assess the non-neuropathic or neuropathic pain and describe the different qualities of pain and related symptoms. It has 0 to 10 scale, with 0 begin no pain and 10 begin worst pain.
Short Form McGill Pain Questionnaire | 8 weeks
  Short Form McGill Pain Questionnaire is used to assess the non-neuropathic or neuropathic pain and describe the different qualities of pain and related symptoms. It has 0 to 10 scale, with 0 begin no pain and 10 begin worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid O Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Wazir Memorial Hospital, Toba Tek Singh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman EL, Callaghan BC, Pop-Busui R, Zochodne DW, Wright DE, Bennett DL, Bril V, Russell JW, Viswanathan V. Diabetic neuropathy. Nat Rev Dis Primers. 2019 Jun 13;5(1):41. doi: 10.1038/s41572-019-0092-1. PMID 31197153
- [Background] Kessler NJ, Lockard MM, Fischer J. Whole body vibration improves symptoms of diabetic peripheral neuropathy. J Bodyw Mov Ther. 2020 Apr;24(2):1-3. doi: 10.1016/j.jbmt.2020.01.004. Epub 2020 Feb 11. PMID 32507132
- [Background] Rippetoe J, Wang H, James SA, Dionne C, Block B, Beckner M. Improvement of Gait after 4 Weeks of Wearable Focal Muscle Vibration Therapy for Individuals with Diabetic Peripheral Neuropathy. J Clin Med. 2020 Nov 22;9(11):3767. doi: 10.3390/jcm9113767. PMID 33266464
- [Background] Chandrashekhar R, Wang H, Dionne C, James S, Burzycki J. Wearable Focal Muscle Vibration on Pain, Balance, Mobility, and Sensation in Individuals with Diabetic Peripheral Neuropathy: A Pilot Study. Int J Environ Res Public Health. 2021 Mar 2;18(5):2415. doi: 10.3390/ijerph18052415. PMID 33801216